CLINICAL TRIAL: NCT02713165
Title: Effects of Adding Raisins to the American Diet on Fecal Microbiota Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Sun-Maid Growers of California (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201500607
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Inflammation
Keywords: Gut Microbiota
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raisins Enhanced Diet (Experimental): Participants will be provide with a Raisin Enhanced Diet over a short term period of time.
  Interventions: Other: Raisins

INTERVENTIONS:
Other: Raisins — Participants will consume 84g of raisins per day for 14 days.
  Other Names: Sun-Maid California Raisins

SUMMARY:
Raisins contain a significant amount of dietary fiber and polyphenolic compounds that represent an important substrate for microbiota fermentation which generates potentially beneficial end products, such as short-chain fatty acids. The mammalian gut contains a phylogenetically as well as functionally diverse microbiota that contributes to host physiology. To date, little is known about how increased raisin intake affects human gut microbiota composition.

This research study will assess the effects of adding raisins to the diet of healthy adults on the bacteria from feces of human subjects and resulting self-reported GI symptoms as well as markers of immune function. The hypothesis is that by adding raisins to the diet this will result in changes in gut microbiota. Furthermore, the changes in microbiota will largely be beneficial, as evaluated by an increase in butyrate producers and bacteria associated with anti-inflammatory properties.

DETAILED DESCRIPTION:
The research study design is a 14 day international focus on increasing raising intake. Participants will be provided with a commercial raisin product for a 14 day period. Participants will consume 2 servings/day (84g of raisins). While participants will be told to substitute raisins for other diet ingredients, they will be free to choose what to substitute according to their preferences. Participants will keep daily food records and will be told that raisin consumption will be monitored in their fecal samples (qPCR). Fecal samples will be collected before the start (Day1), during (Day5-7) and at the end (Day 12-14) of the intervention using a stool collection kit (Sigma). Participants will complete a GI health questionnaire on a weekly basis to determine tolerance to increased raisin intake.

ELIGIBILITY:
Inclusion Criteria:

* Good Health
* No systemic antibiotics during the preceding two months
* No medication suppressing immune function
* Willingness to provide basic demographic as well as medical history data

Exclusion Criteria:

* Gastric Ulcers
* Inflammatory Bowel Disease (IBD) or Irritable Bowel Syndrome (IBS)
* Chronic constipation/diarrhea
* Body Mass Index (BMI) > 30
* Dietary restrictions that prevent legume intake
* Currently on any medication that can affect GI transit time
* Consumption of >3 servings/week of raisins BEFORE study begins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in diversity of gut microbiota 16S rRNA gene sequences with regard to time. | Change in Baseline (Day 1), Day 9, and Day 14
  Compare the overall gut microbial diversity of individual subjects before and after the implementation of a controlled and observed diet of raisins, using 16S ribosomal RNA (rRNA) sequencing of fecal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Mai, PhD, MPH, Principal Investigator — Associate Professor
Locations (1):
- Emerging Pathogens Institiute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wijayabahu AT, Waugh SG, Ukhanova M, Mai V. Dietary raisin intake has limited effect on gut microbiota composition in adult volunteers. Nutr J. 2019 Mar 7;18(1):14. doi: 10.1186/s12937-019-0439-1. PMID 30845997